CLINICAL TRIAL: NCT05779696
Title: Understanding and Identifying the Potential of Artificial Intelligence Powered Digital Physical Activity and Lifestyle Interventions Among People From Ethnic Minority Groups: a Mixed Methods Study
Brief Title: Artificial Intelligence and Physical Activity Among People From Ethnic Minority Groups
Acronym: AI-ACTIV-E
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Responsible Party: Principal Investigator, Tom Wilkinson, Research Fellow, University of Leicester
Other Study IDs: 39522
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Physical Inactivity
Keywords: Physical activity; Artificial intelligence; Ethnic health
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: We will recruit a diverse range of participants to take part and therefore have a limited inclusion/exclusion criteria. Participants must be over 18 years old and be able to a computer/mobile device to access the survey or video conference software (Zoom, as used by the Centre of Ethnic Health Research). Participants can come from a range of cultural communities and religious groups. Participants do not need to have any prior knowledge to participate in the virtual focus groups or the survey.
  Interventions: Other: No-intervention

INTERVENTIONS:
Other: No-intervention — This is a non-intervention study.

SUMMARY:
Despite the high interest in physical activity, many individuals lack the necessary experience in being active and therefore have low levels of knowledge and confidence to become and stay active. For effective lifestyle changes to occur, information must be tailored to the individual's health, goals, motivations, and overall ability. Lifestyle interventions, for example those designed to increase physical activity, are only effective when adapted to the physical, social, and psychological needs of the patient and progressed at rate appropriate for their development by specialist health professional. In the context of ethnic minority health, information must also be culturally adapted, sensitive to religious needs, and accessible to those where English is not proficient. Behavioural digital health interventions have been moderately successful in increasing physical activity, although opportunities for further improvement remain to be discussed. New technologies involving the use of artificial intelligence (AI) are growing, and allow the dissemination of individualised and tailored advice and information. Whilst a few AI-driven physical activity-based applications exist, they are not widely used, particularly amongst people from ethnic minority groups where both physical activity and digital health literacy is poor. Research has identified that whilst many people would be receptive to using health chatbots, hesitancy regarding this technology is likely to compromise engagement. In particular, user perspectives, motivation and capabilities need to be taken into account when developing and assessing the effectiveness of health chatbots. Guidance suggests that developing health chatbots should focus on issues of digital literacy, linguistic and cultural issues, privacy concerns, and personalization. As such, any development needs to involve user-driven co-creation techniques and involving community partners to increase the probability that it will ultimately be effective.

Aims

Aim 1 Gain a new understanding of barriers and facilitators to digital physical activity interventions and AI-delivered healthcare in people from ethnic minority groups through an online survey

Aim 2 To conduct a series of focus groups to explore participants understanding and identifying barriers and facilitators to digital physical activity interventions. In particular to:

i)Better understand general barriers and facilitators (focus on access and provision of education, and physical, environmental, cultural and psycho-social barriers) to physical activity; ii)Explore current and future usage of digital-based resources to facilitate physical activity behaviour; iii)Investigate views of use of AI in digital-based healthcare applications (e.g., trust in such applications)

ELIGIBILITY:
Inclusion

* Participants must be over 18 years old;
* Participants must be able to a computer/mobile device to access the survey or video conference software (Zoom, as used by the Centre of Ethnic Health Research)
* Participants can come from a range of cultural communities and religious groups;
* Participants do not need to have any prior knowledge to participate in the virtual focus groups or the survey.

Exclusion

- No specific exclusion criteria.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We aim to recruit a range of people from different ethnic minority groups - we are interested in a diverse sample of participants with a wide-ranging view on the use of digital-health based interventions and AI.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Feelings towards chatbots and artificial intelligence | 12 months
  Bespoke questions via online survey. Questions answered on a Likert scale between 1 and 7; with 1 being 'disagree completely' and 7 being 'agree completely'

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Wilkinson, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared.

REFERENCES:
- See also: Webpage for study — https://ethnichealthresearch.org.uk/ai-activ-e/